CLINICAL TRIAL: NCT01474512
Title: A Multicenter Study With a Randomized, Double-Blind, Placebo-Controlled Induction Dosing Period Followed by a Randomized Maintenance Dosing Period and a Long- Term Extension Period to Evaluate the Efficacy and Safety of LY2439821 in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Phase 3 Study in Participants With Moderate to Severe Psoriasis
Acronym: UNCOVER-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12972; I1F-MC-RHAZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-01-18

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 80 milligrams (mg) Ixekizumab Dosing Regimen 1 (Q2W) (Experimental): Administered as two 80-mg subcutaneous (SC) injections at Week 0, then one 80-mg SC injection per Dosing Regimen 1 [every 2 weeks (Q2W)] up to and including Week 10. At Week 12, arm is re-randomized to placebo, Dosing Regimen 2 [every 4 weeks (Q4W)] or Dosing Regimen 3 [every 12 weeks Q12W)].
  Interventions: Drug: 80 mg Ixekizumab Dosing Regimens 1, 2, and 3
- 80 mg Ixekizumab Dosing Regimen 2 (Q4W) (Experimental): Administered as two 80-mg SC injections at Week 0, then one 80-mg SC injection per Dosing Regimen 2 (Q4W) up to and including Week 10. At Week 12, arm is re-randomized to placebo, Dosing Regimen 2 (Q4W) or Dosing Regimen 3 (Q12W).
  Interventions: Drug: 80 mg Ixekizumab Dosing Regimens 1, 2, and 3
- 80 mg Ixekizumab Dosing Regimen 3 (Q12W) (Experimental): Dosing Regimen 3 (Q12W) is not used until Week 12. At Week 12, participants who were re-randomized to this arm were administered one 80-mg SC injection Q12W.
  Interventions: Drug: 80 mg Ixekizumab Dosing Regimens 1, 2, and 3
- Placebo (Placebo Comparator): Administered as 2 SC injections at Week 0, then 1 SC injection per Dosing Regimen 1 (Q2W) up to and including Week 10. At Week 12, arm is re-randomized to placebo or Dosing Regimen 2 (Q4W).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 80 mg Ixekizumab Dosing Regimens 1, 2, and 3 — Administered SC
  Other Names: LY2439821
  Arms: 80 mg Ixekizumab Dosing Regimen 2 (Q4W); 80 mg Ixekizumab Dosing Regimen 3 (Q12W); 80 milligrams (mg) Ixekizumab Dosing Regimen 1 (Q2W)
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of LY2439821 compared to placebo in participants with moderate to severe, chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque psoriasis based on a confirmed diagnosis of chronic psoriasis vulgaris for at least 6 months prior to randomization
* At least 10% Body Surface Area (BSA) of Psoriasis at screening and at randomization
* Static Physician Global Assessment (sPGA) score of at least 3 and Psoriasis Area and Severity Index (PASI) score of at least 12 at screening and at randomization
* Candidate for phototherapy and/or systemic therapy
* Men must agree to use a reliable method of birth control during the study
* Women must agree to use birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment

Exclusion Criteria:

* Pustular, erythrodermic, and/or guttate forms of psoriasis
* History of drug-induced psoriasis
* Clinically significant flare of psoriasis during the 12 weeks prior to randomization
* Concurrent or recent use of any biologic agent
* Received systemic psoriasis therapy [such as psoralen and ultraviolet A (PUVA) light therapy] or phototherapy within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks prior to randomization
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to randomization and during the study
* Have participated in any study with interleukin (IL)-17 antagonists, including LY2439821
* Serious disorder or illness other than plaque psoriasis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1296 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (104):
- United States (34):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bakersfield, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremont, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miramar, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ormond Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pinellas Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington Heights, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Owensboro, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnston, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellingham, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- Australia (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benowa, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloogabba, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carlton, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremantle, Western Australia
- Canada (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surrey, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moncton, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ajax, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrie, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newmarket, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond Hill, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Windsor, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hellerup
- Germany (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darmstadt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mahlow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quedlinburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuppertal
- Hungary (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miskolc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szombathely
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
- Japan (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salford, Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scunthorpe, North Lincolnshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dundee, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuneaton, Warwickshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lanarkshire

REFERENCES:
- [Derived] Egeberg A, Hawkes JE, Somani N, Burge R, See K, Gallo G, McKean-Matthews M, Gooderham M, Han G, Armstrong A. Sustained Improvements in Clinical and Patient-Reported Outcomes and Quality of Life Through 5 Years Among Ixekizumab-Treated Patients with Complete Clearance of Scalp Psoriasis by Week 60. Dermatol Ther (Heidelb). 2024 Apr;14(4):1007-1018. doi: 10.1007/s13555-024-01147-7. Epub 2024 Apr 22. PMID 38647975
- [Derived] Kirkham BW, Egeberg A, Behrens F, Pinter A, Merola JF, Holzkamper T, Gallo G, Ng KJ, Bolce R, Schuster C, Nash P, Puig L. A Comprehensive Review of Ixekizumab Efficacy in Nail Psoriasis from Clinical Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Rheumatol Ther. 2023 Oct;10(5):1127-1146. doi: 10.1007/s40744-023-00553-1. Epub 2023 Jul 3. PMID 37400681
- [Derived] Elewski BE, Blauvelt A, Gallo G, Wolf E, McKean-Matthews M, Burge R, Merola JF, Gottlieb AB, Guenther LC. Simultaneous Nail and Skin Clearance in Ixekizumab Head-to-Head Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Dermatol Ther (Heidelb). 2022 Apr;12(4):911-920. doi: 10.1007/s13555-022-00704-2. Epub 2022 Mar 13. PMID 35279805
- [Derived] Leonardi C, Reich K, Foley P, Torii H, Gerdes S, Guenther L, Gooderham M, Ferris LK, Griffiths CEM, ElMaraghy H, Crane H, Patel H, Burge R, Gallo G, Shrom D, Leung A, Lin CY, Papp K. Efficacy and Safety of Ixekizumab Through 5 Years in Moderate-to-Severe Psoriasis: Long-Term Results from the UNCOVER-1 and UNCOVER-2 Phase-3 Randomized Controlled Trials. Dermatol Ther (Heidelb). 2020 Jun;10(3):431-447. doi: 10.1007/s13555-020-00367-x. Epub 2020 Mar 21. PMID 32200512
- [Derived] Gordon KB, Blauvelt A, Papp KA, Langley RG, Luger T, Ohtsuki M, Reich K, Amato D, Ball SG, Braun DK, Cameron GS, Erickson J, Konrad RJ, Muram TM, Nickoloff BJ, Osuntokun OO, Secrest RJ, Zhao F, Mallbris L, Leonardi CL; UNCOVER-1 Study Group; UNCOVER-2 Study Group; UNCOVER-3 Study Group. Phase 3 Trials of Ixekizumab in Moderate-to-Severe Plaque Psoriasis. N Engl J Med. 2016 Jul 28;375(4):345-56. doi: 10.1056/NEJMoa1512711. Epub 2016 Jun 8. PMID 27299809
- [Derived] Armstrong AW, Lynde CW, McBride SR, Stahle M, Edson-Heredia E, Zhu B, Amato D, Nikai E, Yang FE, Gordon KB. Effect of Ixekizumab Treatment on Work Productivity for Patients With Moderate-to-Severe Plaque Psoriasis: Analysis of Results From 3 Randomized Phase 3 Clinical Trials. JAMA Dermatol. 2016 Jun 1;152(6):661-9. doi: 10.1001/jamadermatol.2016.0269. PMID 26953848

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Induction Period (Week 0 to 12), Maintenance Period (Week 12 to 60); Long term Extension (Week 60 to 264) and Post treatment ( last treatment visit (week 264), or Early Termination Visit (ETV) up to a minimum of 12 weeks following that visit.
Pre-assignment Details: Participants received Ixekizumab (ixe) as responders (Resp, sPGA 0/1) in Induction (IND) re-randomized to receive ixe Q4W, Q12W or placebo (PBO) in Maintenance (MAIN) [Primary Population (Pop)]. In MAIN, non-responders (Non-Resp, sPGA >1) in IND received ixe Q4W, PBO Resp in IND received PBO (Secondary Pop). Ixe or PBO continued to end of study.
Groups:
- Placebo- Induction Period: Placebo was administered as 2 subcutaneous (SC) injections at week 0 then 1 PBO (SC) injection every 2 weeks (Q2W) up to Week 10.
- Ixe Q4W - Induction Period: 160 milligrams (mg) ixe was administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection every 4 weeks (Q4W). Placebo was administered as 1 SC injection at Weeks 2, 6, and 10.
- Ixe Q2W - Induction Period: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q2W at Weeks 2, 4, 6, 8, and 10.
- Ixe/Placebo- Maintenance Period Primary Pop: Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56.
- Ixe/Ixe Q12W - Maintenance Period Primary Pop: Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection every 12 weeks (Q12W) up to and including Week 56. Pbo injection was given in between doses Q4W to maintain blindness.
- Ixe/Ixe Q4W - Maintenance Period Primary Pop: Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Placebo Resp/Placebo - Maintenance Period Secondary Pop: Participants who received Placebo during the Induction Period (Weeks 0 to 10) and classified as responders and were administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56.
- Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop: Participants who received placebo in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 160 mg ixe as 2 SC injections at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q4W Non-Resp/Ixe Q4W- Maintenance Period Secondary Pop: Participants who received 80 mg ixe Q4W in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop: Participants who received 80 mg ixe Q2W in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q4W - Maintenance Period Relapsed Population: Participants who relapsed during maintenance period prior to long term received, Ixe 80 mg as 1 SC injection Q4W for the remainder of the study to evaluate whether the response observed earlier could be regained on treatment with a higher dose.
- Placebo Long-Term Extension (LTE): Participants who received placebo at the start of the long-term extension period and remained on placebo. Participants who received placebo at the start of long-term extension period (Week 60) then switched to Ixe.
- Ixe Long-Term Extension: Participants who received 80 mg ixe in all dosing regimens at the start of the long-term extension period from Week 60 to Week 264.
- Total Ixe Long-Term Extension: Participants who received at least 1 dose of 80 mg ixe in all dosing regimens during the long-term extension period from Week 60 to Week 264, including those who have switched from PBO to Ixe in long-term extension (LTE) period.
- Placebo Post-Treatment Follow-Up: Participants who received PBO prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe Q12W Post-Treatment Follow-Up: Participants who received 80 mg ixe 1 SC injection Q12W prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe Q4W Post-Treatment Follow-Up: Participants who received 80 mg ixe Q4W prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe Q2W Post-Treatment Follow-Up: Participants who received 80 mg ixe Q2W prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
Period: Induction Period
Arm/Group | Placebo- Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W Non-Resp/Ixe Q4W- Maintenance Period Secondary Pop | Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop | Ixe Q4W - Maintenance Period Relapsed Population | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 431 | 432 | 433 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Study Drug | 431 | 432 | 433 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 407 | 408 | 415 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 24 | 24 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 10 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Placebo- Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W Non-Resp/Ixe Q4W- Maintenance Period Secondary Pop | Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop | Ixe Q4W - Maintenance Period Relapsed Population | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 0 | 0 | 0 | 226 | 227 (One participant withdrew end of Induction but re-randomized and treated with maintenance dose ixe.) | 229 | 16 | 391 | 78 | 62 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Study Drug | 0 | 0 | 0 | 226 | 227 | 229 | 16 | 391 | 78 | 62 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Relapsed Population Received Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 348 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Relapsed Population Completers | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 321 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 24 | 108 | 177 | 6 | 350 | 62 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 202 | 119 | 52 | 10 | 41 | 16 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Relapsed (sPGA ≥3) | 0 | 0 | 0 | 186 | 111 | 39 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 2 | 7 | 0 | 19 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6 | 2 | 3 | 1 | 6 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Relapse | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 11 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Treated but Discontinued in Induction | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Extension Period
Arm/Group | Placebo- Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W Non-Resp/Ixe Q4W- Maintenance Period Secondary Pop | Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop | Ixe Q4W - Maintenance Period Relapsed Population | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 (9 participants did not start the long-term extension period.) | 1054 (Participants received Ixe alone at the start of long-term extension.) | 1075 (Participants received Ixe in all dosing regimens, including participants who switched PBO to Ixe.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 836 | 855 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 218 | 220 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 61 | 61 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 57 | 58 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 25 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 24 | 25 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 21 | 0 | 0 | 0 | 0
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 0 | 0 | 0 | 0
Not completed — Parent/Caregiver Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Switched From PBO to Ixe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post-Treatment Follow-Up
Arm/Group | Placebo- Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W Non-Resp/Ixe Q4W- Maintenance Period Secondary Pop | Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop | Ixe Q4W - Maintenance Period Relapsed Population | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 (Includes participants who started the post treatment follow-up period.) | 25 (Includes participants who started the post treatment follow-up period.) | 700 (Includes participants who started the post treatment follow-up period.) | 285 (Includes participants who started the post treatment follow-up period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 544 | 239
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 8 | 156 | 46
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 58 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 36 | 17
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 31 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Not completed — Parent/Caregiver Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Placebo administered as 2 SC injections Q2W up to Week 10.
- Ixe Q4W: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q4W.
- Ixe Q2W: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q2W up to Week 10.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W | Total
Number analyzed (Participants) | 431 | 432 | 433 | 1296
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.40) | 45.6 (12.95) | 45.1 (12.40) | 45.7 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 143 | 142 | 413
  Male | 303 | 289 | 291 | 883
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 77 | 69 | 66 | 212
  Romania | 8 | 3 | 2 | 13
  Hungary | 23 | 17 | 26 | 66
  United States | 146 | 156 | 159 | 461
  Japan | 13 | 12 | 8 | 33
  Denmark | 4 | 4 | 8 | 16
  Poland | 43 | 41 | 55 | 139
  Italy | 3 | 2 | 1 | 6
  United Kingdom | 7 | 7 | 7 | 21
  Australia | 19 | 15 | 8 | 42
  Germany | 88 | 106 | 93 | 287
Static Physician Global Assessment (sPGA) [Count of Participants; unit: Participants] — The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe).
  Participants
    sPGA=3 | 204 | 197 | 231 | 632
    sPGA=4, 5 | 227 | 235 | 202 | 664
Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — PASI combines body surface involvement in 4 regions (head, trunk, arms, and legs), percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for final PASI, calculated as: sum of severity parameters for each region*area score*weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Scores range from 0 (no Ps) to 72 (the most severe disease).
  units on a scale | 20.32 (8.641) | 20.03 (7.304) | 20.09 (7.992) | 20.15 (7.992)
Itch Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10 (worst itch imaginable). Overall severity of a participant's itching from psoriasis (Ps) is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
  units on a scale | 7.0 (2.58) | 7.0 (2.50) | 7.2 (2.39) | 7.1 (2.49)
Dermatology-Specific Quality of Life Index (DLQI) Score [Mean (Standard Deviation); unit: units on a scale] — DLQI is a participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include 0 (not at all), 1 (a little), 2 (a lot), and 3 (very much) and unanswered ("not relevant") responses were scored as "0." Total scores range from 0 to 30, with higher score indicating greater quality of life is impairment.
  units on a scale | 12.8 (7.11) | 13.2 (7.02) | 13.4 (7.02) | 13.1 (7.05)
Nail Psoriasis Severity Index (NAPSI) [Mean (Standard Deviation); unit: units on a scale] — The NAPSI is a numeric, reproducible, objective tool to evaluate the severity of fingernail bed Ps and fingernail matrix Ps. Each fingernail is given a score for fingernail bed Ps and fingernail matrix Ps, each with scores of 0 (none) to 4 (Ps in all 4 quadrants) depending on the features of each fingernail bed and fingernail matrix Ps.The NAPSI score of a fingernail is the sum of scores in fingernail bed and fingernail matrix from each quadrant (maximum of 8). The sum of all fingernails equals the total NAPSI score with a range from 0 to 80. Higher scores indicated more severe psoriasis. Population: ITT population: all randomized participants analyzed according to the treatment to which they are assigned; and had fingernail Ps at baseline.
  units on a scale
    number analyzed (Participants) | 283 | 281 | 283 | 847
    (all) | 26.9 (20.492) | 24.12 (18.243) | 24.64 (18.916) | 24.95 (19.238)
Percent of Body Surface Area (BSA) involvement of Ps [Mean (Standard Deviation); unit: percent of body surface] — BSA is a physician rating of the percentage of involvement of Ps for each participant. BSA is assessed on a continuous scale from 0% (no involvement) to 100% (full involvement), where 1% corresponds to the size of the participants hand (includes the palm, fingers and thumb).
  percent of body surface | 27.4 (17.77) | 27.4 (16.20) | 28.2 (17.83) | 27.7 (17.27)
Psoriasis Scalp Severity Index (PSSI) [Mean (Standard Deviation); unit: units on a scale] — The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total scores range from 0 to 72, with lower scores indicating less severity. Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and had scalp Ps at baseline.
  units on a scale
    number analyzed (Participants) | 393 | 413 | 393 | 1199
    (all) | 21.8 (15.70) | 19.9 (14.83) | 21.1 (14.69) | 20.9 (15.08)
Quick Inventory of Depressive Symptomatology-Self Reported 16 Items (QIDS-SR16) [Mean (Standard Deviation); unit: units on a scale] — QIDS-SR16 is a participant-administered, 16-item instrument to assess the existence and severity of depression symptoms. A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days and rate each on a 4-point scale: 0 (best) to 3 (worst). The sum of the 16 items corresponding to 9 depression domains (sad mood, concentration, self-criticism, suicidal ideation, interest, energy, sleep disturbance, change in appetite/weight, and psychomotor agitation/retardation) to give a total scores range from 0 to 27, higher scores indicate greater severity. Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned, and had results at the specified time points, LOCF.
  units on a scale
    number analyzed (Participants) | 430 | 431 | 431 | 1292
    (all) | 4.7 (4.34) | 5.0 (4.34) | 4.5 (4.09) | 4.8 (4.26)
Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO) [Mean (Standard Deviation); unit: units on a scale] — WPAI-PSO is a self-administered, 6-item instrument used to assess the impact of Ps on productivity impairment within the past 7 days. WPAI-PSO has 4 domains: absenteeism, presenteeism (reduced productivity at work), an overall work impairment score and impairment in daily activities performed outside work. Four scores are derived as percentages: absenteeism, presenteeism (reduced productivity while at work), overall work impairment (absenteeism and presenteeism), and impairment in activities performed outside of work. Percentage = each score * 100. Greater scores indicate greater impairment. Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned, and had results at specified time points, last observation carried forward (LOCF).
  units on a scale
    Absenteeism: number analyzed (Participants) | 281 | 287 | 290 | 858
    Absenteeism | 4.5 (17.07) | 4.0 (16.26) | 5.7 (19.41) | 4.7 (17.63)
    Activity Impairment: number analyzed (Participants) | 431 | 429 | 432 | 1292
    Activity Impairment | 31.3 (29.29) | 34.7 (28.83) | 34.2 (28.99) | 33.4 (29.05)
    Presenteeism: number analyzed (Participants) | 297 | 301 | 299 | 897
    Presenteeism | 22.2 (25.85) | 25.2 (27.22) | 22.6 (26.46) | 23.3 (26.53)
    Work Productively Loss: number analyzed (Participants) | 279 | 284 | 288 | 851
    Work Productively Loss | 24.6 (27.90) | 27.0 (27.90) | 24.9 (28.77) | 25.5 (28.18)
Medical Outcomes Study 36-Item Short Form (SF36) Physical component (PCS) and Mental Component (MCS) [Mean (Standard Deviation); unit: units on a scale] — The SF-36 is a self-reported instrument that measures the participant's health status during the previous 7 days. It comprises 36-items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped in the PCS and MCS scores. Scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and with results at the specified time points, LOCF.
  units on a scale
    PCS: number analyzed (Participants) | 428 | 428 | 432 | 1288
    PCS | 46.92 (9.769) | 47.34 (9.169) | 46.58 (9.146) | 46.95 (9.363)
    MCS: number analyzed (Participants) | 428 | 428 | 432 | 1288
    MCS | 48.77 (11.182) | 47.46 (11.655) | 47.94 (11.535) | 48.05 (11.463)
Patient's Global Assessment of Disease Severity (PatGA) [Mean (Standard Deviation); unit: units on a scale] — The PatGA is a single-item self-reported instrument asking the participant to rate severity of their psoriasis "today" by circling a number on a 0 to 5 numeric rating scale from 0 (Clear = no psoriasis) to 5 (Severe = the worst their psoriasis has ever been). Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and with at least 1 post-baseline PatGA measurement.
  units on a scale
    number analyzed (Participants) | 431 | 430 | 430 | 1291
    (all) | 4.1 (0.95) | 4.1 (0.88) | 4.1 (0.94) | 4.1 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Static Physician Global Assessment (sPGA) of 0 or 1 (Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Ps Measure: sPGA)
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Time Frame: Week 12
Population: Intent to Treat (ITT) Population: all randomized participants analyzed according to the treatment to which they were assigned. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo was administered as 2 SC injections Q2W (Weeks 2, 4, 6, 8, and 10).
- Ixe Q4W: 160 mg ixe was administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q4W (Weeks 4 and 8).
- Ixe Q2W: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 431 | 432 | 433
percentage of participants | 3.2 | 76.4 | 81.8
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic Regression analysis included treatment, geographic region, previous non-biologic systemic therapy and baseline weight category as factors
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants Achieving ≥75% Improvement in Ps Area and Severity Index (PASI75) (Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Psoriasis Measure: PASI)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease). Participants achieving PASI75 were defined as having an improvement of ≥75% in the PASI score compared to baseline.
Time Frame: Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they were assigned. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 431 | 432 | 433
percentage of participants | 3.9 | 82.6 | 89.1
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Achieving an sPGA of 0 (Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Ps Measure: sPGA)
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe).
Time Frame: Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 431 | 432 | 433
percentage of participants | 0.0 | 34.5 | 37.0
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Fisher Exact; Due to the zero count in placebo group, p-values from Logistic Regression were not obtainable, therefore the p-value is from Fisher's exact test
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Fisher Exact; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving PASI 90% (PASI90) or 100% (PASI100) (Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Ps Measure: PASI)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease). Participants achieving PASI90 or PASI100 were defined as having an improvement of ≥90% or of 100% respectively in PASI scores compared to baseline.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 431 | 432 | 433
percentage of participants
  PASI90 | 0.5 | 64.6 | 70.9
  PASI100 | 0.0 | 33.6 | 35.3
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for PASI90; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for PASI90; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for PASI100; Due to the zero count in placebo group, p-values from Logistic Regression were not obtainable; therefore the p-value is from Fisher's exact test
Statistical Analysis 4: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for PASI100; [statistical method as in outcome 4, analysis 3]

5. Secondary Outcome: Percentage of Participants Maintaining sPGA 0 or 1 After Re-Randomization at Start of Maintenance Dosing Period
Description: as for outcome 3
Time Frame: Week 60
Population: Maintenance Period Primary Population (MPPP): all randomized participants from Period 2 who achieved sPGA (0, 1), were re-randomized at Week 12 and who received at least 1 dose of study treatment Period 3. Participants did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Groups:
- Ixe/Placebo: Participants who received ixe (Q2W or Q4W) in Induction Period who were re-randomized at Week 12 and administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56 (Maintenance Period).
- Ixe/Q12W: Participants who received ixe (Q2W or Q4W) in Induction Period who were re-randomized at Week 12 and were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection Q12W up to and including Week 56 (Maintenance Period).
- Ixe/Q4W: Participants who received ixe (Q2W or Q4W) in Induction Period who were re-randomized at Week 12 and were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56 (Maintenance Period).
Arm/Group | Ixe/Placebo | Ixe/Q12W | Ixe/Q4W
Number analyzed (Participants) | 226 | 227 | 229
percentage of participants | 7.5 | 37.4 | 72.9
Statistical Analysis 1: Comparison: Ixe/Placebo vs Ixe/Q12W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic Regression analysis included treatment and baseline weight category as factors
Statistical Analysis 2: Comparison: Ixe/Placebo vs Ixe/Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic Regression analysis included treatment and baseline weight category as factors

6. Secondary Outcome: Percentage of Participants With Itch Numeric Rating Scale (Itch NRS) Score ≥4 Point Reduction From Baseline
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10 (worst itch imaginable). Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and had an Itch NRS score ≥4 at baseline. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 374 | 379 | 391
percentage of participants | 15.5 | 80.5 | 85.9
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Dermatology-Specific Quality of Life Index (DLQI) Score
Description: DLQI is a participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include 0 (not at all), 1 (a little), 2 (a lot), and 3 (very much) and unanswered ("not relevant") responses were scored as "0." Total scores range from 0 to 30, with higher score indicating greater quality of life is impairment. A 5-point change from baseline is considered clinically relevant. Least squares (LS) mean change from baseline was calculated using mixed model repeated measures (MMRM).
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and who had at least 1 post-baseline DLQI measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 421 | 421 | 427
units on a scale | -1.0 (0.27) | -10.7 (0.27) | -11.1 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — LS mean and P-value were calculated using MMRM with baseline score as a covariate, treatment, geographic region, previous non-biologic systemic therapy, baseline weight category, visit and treatment-by-visit interaction as fixed effects
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI)
Description: The NAPSI is a numeric, reproducible, objective tool for evaluation of fingernail Ps. This scale is used to evaluate the severity of fingernail bed Ps and fingernail matrix Ps by area of involvement in the fingernail unit. The fingernail is divided with imaginary horizontal and longitudinal lines into quadrants. Each fingernail is given a score for fingernail bed Ps 0 (none) to 4 (Ps in 4 quadrants of the fingernail) and fingernail matrix Ps 0 (none) to 4 (Ps in 4 quadrants of the matrix), depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed or matrix Ps in each quadrant. The NAPSI score of a fingernail is the sum of scores in fingernail bed and fingernail matrix from each quadrant (maximum of 8). Each fingernail is evaluated, then the sum of all fingernails equals the total NAPSI score with a range from 0 to 80 with higher scores indicating more severe psoriasis. LS mean change from baseline was calculated using MMRM.
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and had fingernail Ps at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 280 | 276 | 279
units on a scale | 2.17 (0.672) | -7.19 (0.671) | -7.24 (0.657)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]

9. Secondary Outcome: Percent of Body Surface Area (BSA) Involvement of Ps
Description: BSA is a physician rating of the percentage of involvement of Ps for each participant. BSA is assessed on a continuous scale from 0% (no involvement) to 100% (full involvement), where 1% corresponds to the size of the participants hand (includes the palm, fingers and thumb). Total BSA is the sum of handprints from the affected areas. LS mean change from baseline was calculated using MMRM.
Time Frame: Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and had at least 1 post-baseline BSA measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 426 | 425 | 428
percentage of body surface | 1.3 (0.67) | -21.4 (0.67) | -22.4 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in Psoriasis Scalp Severity Index (PSSI)
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total scores range from 0 to 72, with lower scores indicating less severity. LS mean change from baseline was calculated using MMRM.
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and had scalp Ps at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 393 | 413 | 393
units on a scale | -1.8 (0.53) | -18.3 (0.52) | -19.2 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]

11. Secondary Outcome: Change From Baseline in All Scores of the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO) Quality of Life and Outcome Assessments. Measures: Participant Reported Outcomes (PRO)
Description: WPAI-PSO is a participant administered, 6-item instrument used to assess the impact of Ps on the productivity impairment within the past 7 days. WPAI-PSO has 4 domains: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score, and impairment in daily activities performed outside of work. Four scores are derived as percentages: absenteeism, presenteeism (reduced productivity while at work), overall work impairment (absenteeism and presenteeism), and impairment in activities performed outside of work. Percentage is calculated as: each score * 100 with greater scores indicating greater impairment. LS mean change from baseline was calculated using analysis of covariance (ANCOVA).
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned, and had results at specified time points, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 420 | 417 | 427
units on a scale
  Absenteeism: number analyzed (Participants) | 253 | 250 | 255
  Absenteeism | 0.2 (0.88) | -3.5 (0.87) | -2.6 (0.84)
  Activity Impairment | 0.8 (1.18) | -24.5 (1.18) | -25.2 (1.15)
  Presenteeism: number analyzed (Participants) | 275 | 273 | 278
  Presenteeism | 0.5 (1.30) | -18.8 (1.28) | -18.3 (1.24)
  Work Productivity Loss: number analyzed (Participants) | 250 | 246 | 252
  Work Productivity Loss | -0.8 (1.40) | -20.6 (1.38) | -19.8 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — The LS Mean and p-values were calculated using an ANCOVA model and included treatment, geographic region, previous non-biologic systemic therapy, baseline weight category, and baseline WPAI value; P-value is for Absenteeism
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value is for absenteeism
Statistical Analysis 3: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value is for activity impairment
Statistical Analysis 4: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value is for activity impairment
Statistical Analysis 5: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value is for presenteeism
Statistical Analysis 6: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value is for presenteeism
Statistical Analysis 7: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value is for work productively loss
Statistical Analysis 8: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value is for work productively loss

12. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptomatology-Self Reported 16 Items (QIDS-SR16)
Description: QIDS-SR16 is a participant-administered, 16-item instrument intended to assess the existence and severity of symptoms of depression. A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days and rate each on a 4-point scale: 0 (best) to 3 (worst). The sum of the 16 items corresponding to 9 depression domains [sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance (initial, middle and late insomnia or hypersomnia), decrease/increase in appetite/weight, and psychomotor agitation/retardation] to give a single total scores range from 0 to 27, with higher scores indicating greater symptom severity. LS mean change from baseline was calculated using ANCOVA.
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned, and had results at the specified time points, LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 421 | 417 | 423
units on a scale | -0.1 (0.17) | -1.0 (0.17) | -1.3 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — LS Mean and p-values were calculated using an ANCOVA model that included treatment, geographic region, previous non-biologic systemic therapy, baseline weight category, and baseline QIDS value in the model
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 12, analysis 1]

13. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-item Short Form Health Survey (SF-36) and Physical Component Summary (PCS) and Mental Component Summary (MCS)
Description: The SF-36 is a self-reported instrument that measures the participant's health status during the previous 7 days. It comprises 36-items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped in the PCS and MCS scores. Scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. LS mean change from baseline was calculated using ANCOVA.
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and with results at the specified time points, LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 418 | 415 | 427
units on a scale
  PCS | -0.1747 (0.4012) | 4.3081 (0.3990) | 4.3159 (0.3878)
  MCS | 0.8729 (0.4638) | 3.7386 (0.4633) | 4.1293 (0.4480)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — The LS Mean and p-values were calculated using an ANCOVA model and included treatment, geographic region, previous non-biologic systemic therapy, baseline weight category, and baseline SF-36 value in the model; P-value is for PCS
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; P-value is for PCS
Statistical Analysis 3: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; P-value is for MCS
Statistical Analysis 4: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; P-value is for MCS

14. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Severity (PatGA)
Description: The PatGA is a single-item self-reported instrument asking the participant to rate the severity of their psoriasis "today" by circling a number on the numeric rating scale from 0 (Clear = no psoriasis) to 5 (Severe = the worst their psoriasis has ever been). LS mean change from baseline calculated using MMRM.
Time Frame: Baseline, Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and with at least 1 post-baseline PatGA measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 424 | 425 | 427
units on a scale | -0.2 (0.06) | -3.1 (0.06) | -3.2 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]

15. Secondary Outcome: Percentage of Participants Achieving Palmoplantar PASI (PPASI) of ≥50% (PPASI50), ≥75% (PPASI75), or 100% (PPASI100) Improvement
Description: The Palmoplantar PASI is a composite score derived from the sum of scores for erythema, induration, and desquamation [scores range from 0 (none) to 4 (very severe) for each] multiplied by the score for the extent of palm and sole area involvement [scores range from 0 (0%) to 6 (90 to100%)], with a total scores range from 0 to 72. Participants achieving PPASI50, PPASI75 or PASI100 were defined as having an improvement of at least 50%, 90%, or of 100%, respectively, in the PPASI scores compared to baseline.
Time Frame: Week 12
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and who had palmoplantar Ps at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 133 | 131 | 140
percentage of participants
  PPASI50 | 35.3 | 84.0 | 82.9
  PPASI75 | 26.3 | 74.8 | 77.1
  PPASI100 | 20.3 | 65.6 | 70.0
Statistical Analysis 1: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for PPASI50; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for PPASI50; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for PPASI75; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for PPASI75; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Ixe Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for PPASI100; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Ixe Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value if for PPASI100; [statistical method as in outcome 1, analysis 1]

16. Secondary Outcome: Pharmacokinetics (PK): Trough Concentration at Steady State (Ctrough ss)
Time Frame: Weeks 12: Day 84 and Week 24: Day 168
Population: ITT Population: all randomized participants analyzed according to the treatment to which they are assigned; and who had Ctrough ss results at specified time points where the concentration met the definition of being a trough concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Groups:
- Ixe Q2W - Induction Period: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
- Ixe Q4W - Induction Period: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q4W (Weeks 4 and 8).
- Ixe Q4W - Maintenance Period: 80 mg ixe administered as 1 SC injection Q4W from Week 12 up to Week 60
- Ixe Q12W - Maintenance Period: 80 mg ixe administered as 1 SC injection Q12W from Week 12 up to Week 60
Arm/Group | Ixe Q2W - Induction Period | Ixe Q4W - Induction Period | Ixe Q4W - Maintenance Period | Ixe Q12W - Maintenance Period
Number analyzed (Participants) | 192 | 215 | 223 | 60
micrograms/milliliter (µg/mL)
  Week 12 | 7.73 (79) | 2.94 (89) | NA (NA) — No Induction Period results available. | NA (NA) — No Induction Period results available.
  Week 24 | NA (NA) — No Maintenance Period results available. | NA (NA) — No Maintenance Period results available. | 2.36 (111) | 0.281 (175)

17. Secondary Outcome: Percentage of Participants With Anti-ixekizumab Antibodies
Description: Percentage of participants with treatment-emergent positive anti-ixekizumab antibodies was summarized by treatment group. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Baseline through Week 12
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixe Q4W | Ixe Q2W
Number analyzed (Participants) | 431 | 432 | 433
percentage of participants | 0.5 | 12.5 | 10.3

ADVERSE EVENTS:
Time Frame: Up to 276 Weeks
Description: All randomized participants who received at least one dose of study drug in induction, maintenance, long-term and post treatment follow-up period. The gender specific events only occurring in male or female participants were adjusted accordingly.
Groups:
- Placebo - Induction Period: Placebo was administered as 2 subcutaneous (SC) injections at week 0 then 1 PBO (SC) injection every 2 weeks (Q2W) up to Week 10.
- Ixe Q4W - Induction Period: 160 mg ixe was administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q4W. Placebo was administered as 1 SC injection at Weeks 2, 6, and 10.
- Ixe Q2W - Induction Period: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q2W up to Weeks 2, 4, 6, 8 and 10.
- Ixe/Ixe Q12W - Maintenance Period Primary Pop: Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection Q12W up to and including Week 56. Pbo injection was given in between doses Q4W to maintain blindness.
- Ixe Q4W Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop: Participants who received 80 mg ixe Q4W in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 80 mg ixe as 1 SC injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q4W - Maintenance Period Relapse Pop: Participants who relapsed (loss of response, sPGA ≥3 during Maintenance Period) were administered 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Placebo Long-Term Extension: Participants who received placebo at the start of the long-term extension period and remained on placebo. Participants who received placebo at the start of long-term extension (Week 60) then switched to Ixe.
- Ixe Long-Term Extension: Participants who received 80 mg ixe in all dosing regimen at the start of the long-term extension period from Week 60 to Week 264
- Total Ixe Long-Term Extension: Participants who received at least 1 dose of 80 mg ixe in all dosing regimens during the long-term extension period from Week 60 to Week 264, including those who have switched from PBO to Ixe in LTE period.
- Ixe Q12W Post-Treatment Follow-Up: Participants who received 80 mg ixe Q12W prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe Q4W Post Treatment Follow-Up: Participants who received 80 mg ixe Q4W prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
Arm/Group | Placebo - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop | Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop | Ixe Q4W - Maintenance Period Relapse Pop | Placebo Long-Term Extension | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Serious Adverse Events (participants affected / at risk) | 5/431 | 12/432 | 7/433 | 7/226 | 11/227 | 14/229 | 0/16 | 24/391 | 8/78 | 3/62 | 11/348 | 1/26 | 134/1054 | 134/1075 | 2/18 | 0/25 | 13/700 | 6/285
Other Adverse Events (participants affected / at risk) | 128/431 | 159/432 | 170/433 | 83/226 | 122/227 | 115/229 | 8/16 | 211/391 | 55/78 | 34/62 | 114/348 | 8/26 | 414/1054 | 414/1075 | 3/18 | 2/25 | 33/700 | 15/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Induction Period (N=431) | Ixe Q4W - Induction Period (N=432) | Ixe Q2W - Induction Period (N=433) | Ixe/Placebo- Maintenance Period Primary Pop (N=226) | Ixe/Ixe Q12W - Maintenance Period Primary Pop (N=227) | Ixe/Ixe Q4W - Maintenance Period Primary Pop (N=229) | Placebo Resp/Placebo - Maintenance Period Secondary Pop (N=16) | Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop (N=391) | Ixe Q4W Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop (N=78) | Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop (N=62) | Ixe Q4W - Maintenance Period Relapse Pop (N=348) | Placebo Long-Term Extension (N=26) | Ixe Long-Term Extension (N=1054) | Total Ixe Long-Term Extension (N=1075) | Placebo Post-Treatment Follow-Up (N=18) | Ixe Q12W Post-Treatment Follow-Up (N=25) | Ixe Q4W Post Treatment Follow-Up (N=700) | Ixe Q2W Post-Treatment Follow-Up (N=285)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital ectopic pancreas (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital pyelocaliectasis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis pharyngeal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 0/107 (0) | 0/11 (0) | 0/323 (0) | 0/332 (0) | 1/5 (1) | 0/15 (0) | 0/215 (0) | 0/78 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac electrophysiologic study (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endoscopic retrograde cholangiopancreatography (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/303 (0) | 0/289 (0) | 0/291 (0) | 0/154 (0) | 0/150 (0) | 0/156 (0) | 0/10 (0) | 0/276 (0) | 0/54 (0) | 0/41 (0) | 0/241 (0) | 0/15 (0) | 1/731 (1) | 1/743 (1) | 0/13 (0) | 0/10 (0) | 0/485 (0) | 0/207 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 0/107 (0) | 0/11 (0) | 1/323 (1) | 1/332 (1) | 0/5 (0) | 0/15 (0) | 0/215 (0) | 0/78 (0)
Hellp syndrome (Pregnancy, puerperium and perinatal conditions) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 0/107 (0) | 0/11 (0) | 0/323 (0) | 0/332 (0) | 0/5 (0) | 0/15 (0) | 1/215 (1) | 0/78 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 0/107 (0) | 0/11 (0) | 0/323 (0) | 0/332 (0) | 0/5 (0) | 0/15 (0) | 1/215 (1) | 0/78 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 0/107 (0) | 0/11 (0) | 1/323 (1) | 1/332 (1) | 0/5 (0) | 0/15 (0) | 0/215 (0) | 0/78 (0)
Endometriosis (Reproductive system and breast disorders) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 0/107 (0) | 0/11 (0) | 1/323 (1) | 1/332 (1) | 0/5 (0) | 0/15 (0) | 0/215 (0) | 0/78 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 1/107 (1) | 0/11 (0) | 2/323 (2) | 2/332 (2) | 0/5 (0) | 0/15 (0) | 0/215 (0) | 0/78 (0)
Rectocele (Reproductive system and breast disorders) | 0/128 (0) | 0/143 (0) | 0/142 (0) | 0/72 (0) | 0/77 (0) | 0/73 (0) | 0/6 (0) | 0/115 (0) | 0/24 (0) | 0/21 (0) | 0/107 (0) | 0/11 (0) | 1/323 (1) | 1/332 (1) | 0/5 (0) | 0/15 (0) | 0/215 (0) | 0/78 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Duodenal sphincterotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia hiatus repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreaticoduodenectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Induction Period (N=431) | Ixe Q4W - Induction Period (N=432) | Ixe Q2W - Induction Period (N=433) | Ixe/Placebo- Maintenance Period Primary Pop (N=226) | Ixe/Ixe Q12W - Maintenance Period Primary Pop (N=227) | Ixe/Ixe Q4W - Maintenance Period Primary Pop (N=229) | Placebo Resp/Placebo - Maintenance Period Secondary Pop (N=16) | Placebo Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop (N=391) | Ixe Q4W Non-Resp/Ixe Q4W - Maintenance Period Secondary Pop (N=78) | Q2W Non-Resp/Q4W - Maintenance Period Secondary Pop (N=62) | Ixe Q4W - Maintenance Period Relapse Pop (N=348) | Placebo Long-Term Extension (N=26) | Ixe Long-Term Extension (N=1054) | Total Ixe Long-Term Extension (N=1075) | Placebo Post-Treatment Follow-Up (N=18) | Ixe Q12W Post-Treatment Follow-Up (N=25) | Ixe Q4W Post Treatment Follow-Up (N=700) | Ixe Q2W Post-Treatment Follow-Up (N=285)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 10 (11) | 9 (11) | 8 (8) | 4 (4) | 8 (8) | 0 (0) | 22 (29) | 1 (1) | 2 (2) | 8 (9) | 1 (1) | 21 (24) | 21 (24) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 18 (24) | 28 (40) | 0 (0) | 3 (3) | 5 (8) | 0 (0) | 13 (15) | 3 (6) | 0 (0) | 2 (9) | 0 (0) | 3 (6) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 5 (5) | 27 (47) | 42 (77) | 2 (2) | 7 (10) | 12 (47) | 0 (0) | 36 (94) | 7 (27) | 2 (10) | 13 (37) | 0 (0) | 27 (302) | 27 (302) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 5 (8) | 0 (0) | 3 (3) | 0 (0) | 14 (14) | 14 (14) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 6 (8) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 2 (3) | 4 (4) | 0 (0) | 17 (22) | 17 (22) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 4 (5) | 8 (8) | 7 (7) | 0 (0) | 7 (7) | 2 (2) | 2 (2) | 3 (4) | 2 (2) | 28 (31) | 28 (31) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 41 (45) | 45 (46) | 49 (57) | 26 (32) | 41 (65) | 51 (71) | 0 (0) | 77 (116) | 19 (25) | 11 (16) | 37 (45) | 4 (7) | 178 (314) | 178 (314) | 0 (0) | 0 (0) | 9 (9) | 1 (1)
Pharyngitis (Infections and infestations) | 6 (6) | 3 (3) | 2 (2) | 5 (5) | 8 (10) | 1 (1) | 1 (1) | 13 (15) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 33 (44) | 33 (44) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 6 (6) | 5 (5) | 7 (8) | 11 (13) | 8 (8) | 1 (1) | 18 (20) | 3 (3) | 2 (3) | 11 (11) | 0 (0) | 46 (56) | 46 (56) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (17) | 20 (20) | 24 (27) | 18 (26) | 20 (22) | 18 (21) | 2 (4) | 53 (76) | 8 (12) | 4 (4) | 18 (21) | 2 (4) | 89 (129) | 89 (129) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 6 (6) | 2 (2) | 3 (3) | 2 (2) | 10 (10) | 0 (0) | 11 (13) | 4 (5) | 2 (4) | 11 (13) | 0 (0) | 31 (48) | 31 (48) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (4) | 9 (12) | 6 (6) | 13 (15) | 13 (16) | 0 (0) | 14 (16) | 8 (10) | 3 (3) | 4 (4) | 1 (1) | 54 (70) | 54 (70) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 4 (6) | 7 (8) | 13 (15) | 6 (6) | 0 (0) | 16 (16) | 1 (1) | 6 (6) | 6 (6) | 0 (0) | 45 (50) | 45 (50) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (4) | 0 (0) | 7 (11) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 17 (18) | 17 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 1 (1) | 2 (3) | 5 (6) | 2 (2) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (14) | 10 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 15 (18) | 16 (21) | 18 (19) | 5 (7) | 16 (19) | 8 (11) | 0 (0) | 20 (26) | 6 (9) | 2 (2) | 6 (11) | 0 (0) | 30 (39) | 30 (39) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 11 (11) | 11 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 7 (7) | 2 (2) | 3 (4) | 3 (3) | 0 (0) | 12 (12) | 5 (6) | 1 (1) | 2 (2) | 0 (0) | 30 (33) | 30 (33) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (10) | 6 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail psoriasis (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) | 3 (3) | 3 (4) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 4 (5) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (12) | 10 (10) | 6 (6) | 3 (4) | 4 (4) | 6 (6) | 1 (1) | 9 (9) | 1 (1) | 2 (3) | 4 (4) | 0 (0) | 12 (13) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 16 (16) | 2 (2) | 4 (4) | 5 (5) | 6 (6) | 2 (2) | 1 (2) | 4 (4) | 2 (2) | 1 (5) | 4 (4) | 0 (0) | 21 (23) | 21 (23) | 0 (0) | 2 (2) | 11 (11) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days